| Statistical<br>Analysis Plan<br>Title: | A Randomised, Double-Blind, Three-Arm, Single Dose, Parallel Study To Compare the Pharmacokinetics, Safety and Immunogenicity of MB02-SP, MB02-DM (Bevacizumab Biosimilar Drugs) and US licenced Avastin® in Healthy Male Volunteers |
|---|---|
| NCT Number: | NCT04408989 |
| Statistical<br>Analysis Plan<br>version date: | Version 1.0, 20 May 2021 |



#### Statistical Analysis Plan (Without PK and Immunogenicity analysis)

# A RANDOMISED, DOUBLE BLIND, THREE-ARM, SINGLE DOSE, PARALLEL STUDY TO COMPARE THE PHARMACOKINETICS, SAFETY AND IMMUNOGENICITY OF MB02-SP, MB02-DM (BEVACIZUMAB BIOSIMILAR DRUGS) AND US LICENCED AVASTIN® IN HEALTHY MALE VOLUNTEERS

Sponsor Protocol No.: MB02-A-06-20 Syneos Health Clinique Inc. Project No.: 7012755

Final Version: 1.0 Date: 26-MAY-2020

Contract Research Organization:
Syneos Health, LLC/ Health UK Limited
1030 Sync Street, Morrisville,
North Carolina 27560,
United States

Sponsor: mAbxience Research S.L. C/ Manuel Pombo Angulo, 28,

4th floor, 28050 Madrid,

Spain

#### CONFIDENTIAL



mAbxience Research S.L.

# **Revision History**

| Version# | Date (DD-Mmm-YYYY) | Document Owner | Revision Summary |
|-----------|--------------------|----------------|------------------|
| Draft 0.1 | 04 May 2021 | | |
| Final 1.0 | 20 May 2021 | | |



# Signature Approvals

I confirm that I have reviewed this document and agree with the content.

| Syneos Health Approval | | |
|---|---|---|
| , Biostatistician II Name, Title Lead Biostatistician | Signature | Date (DD-Mmm-YYYY) |
| , Biostatistician II Name, Title Senior Reviewing Biostatistician | Signature | Date (DD-Mmm-YYYY) |
| , Principal Stat Programmer Name, Title Lead Programmer | Signature | Date (DD-Mmm-YYYY) |
| , Principal Medical Writer Name, Title Lead Medical Writer | Signature | Date (DD-Mmm-YYYY) |
| n | nAbxience Research S.L. | |
| , Medical Advisor Name, Title Spons or Contact | Signature | Date (DD-Mmm-YYYY) |

20 May 2021 (Final 1.0) 



# TABLE OF CONTENTS

| | Rev | vision History | 2 |
|----|------|-------------------------------------------|----|
| | Sign | nature Approvals | 3 |
| | TA | BLE OF CONTENTS | 4 |
| | LIS | T OF ABBREVIATIONS | 6 |
| 1. | | Introduction | 8 |
| 2. | | Study Objectives | 9 |
| | 2.1 | Primary objective | 9 |
| | 2.2 | Secondary objectives | |
| 3. | | Study Design | 10 |
| | 3.1 | General Design | |
| | 3.2 | Study Procedures. | 10 |
| | 3.3 | Drug Administration | 10 |
| | 3.4 | Subject Withdrawal and Replacement | 10 |
| | 3.5 | Determination of Sample Size | |
| | 3.6 | Randomization and Blinding | 11 |
| 4. | | Changes from the Protocol | 13 |
| 5. | | Study Endpoints | |
| | 5.1 | Primary Endpoints | 14 |
| | 5.2 | Secondary Endpoints | 14 |
| 6. | | Analysis Populations | 15 |
| | 6.1 | Safety Population | 15 |
| 7. | | General Aspects for Statistical Analysis | 16 |
| | 7.1 | General Methods | 16 |
| | 7.2 | Summary Statistics: | 16 |
| | 7.3 | Key Definitions | 16 |
| | 7.4 | Missing Data | 17 |
| | 7.5 | Visit Windows | 17 |
| 8. | | Interim Analyses | 18 |
| 9. | | Study Population and Exposure | 19 |
| | 9.1 | Subject Disposition | 19 |
| | 9.2 | Protocol Deviations | |
| | 9.3 | Demographics and Baseline Characteristics | 19 |
| | 9.4 | Medical History | 20 |
| | 9.5 | Prior and Concomitant Medications | 20 |
| | 9.6 | Study Drug Administration | 20 |
| 10 | ). | Safety Analyses | 21 |



mAbxience Research S.L.

| 10. | 1 Physical Examination Findings | 21 |
|------|---------------------------------|----|
| 10.2 | 2 Adverse Events | 21 |
| 10.3 | 3 Laboratory Parameters | 23 |
| 10.4 | 4 Vital Signs | 24 |
| 10.5 | 5 Electrocardiogram | 25 |
| 11. | Percentages and Decimal Places | 26 |
| 12. | Data Handling | 27 |
| | Handling of Missing Data | |
| | Software to be Used. | |
| | Reference List | |



#### LIST OF ABBREVIATIONS

**ADA** Anti-Drug Antibodies

**AE** Adverse Event

anti-HBs Hepatitis B surface antibody

anti HBc Hepatitis B core antibody

**ALP** Alkaline Phosphatase

**ALT** Alanine Aminotransferase

**AST** Aspartate Aminotransferase

**AUC** Area Under the Curve

**BMI** Body Mass Index

**BP** Blood Pressure

BUN Blood urea nitrogen

CI Confidence Interval

CL Total Body Clearance

CTCAE Common Terminology Criteria For Adverse Events

**CR/STBA** Confinement Report and Subjects to be Analyzed Form

**CSR** Clinical Study Report

CV Coefficient of Variation

**ECG** Electrocardiogram

eCRF electronic Case Report Form

**EMA** European Medicines Agency

**EOI** End of Infusion

**EOS** End of Study

**HBsAg** Surface Antigen Of The Hepatitis B Virus

**HCV** Human Hepatitis C Virus

HDL High-Density Lipoprotein

HIV Human Immunodeficiency Virus

HR Heart Rate

INR International Normalised Ratio

IV Intravenous

kg Kilogram



mAbxience Research S.L.

LDL Low-density Lipoprotein

m Meter

Max Maximum

MedDRA Medical Dictionary For Regulatory Activities

mg MilligramMin MinimummL Milliliter

mmHg Millimeters Mercury

NAB Neutralizing Anti-drug antibodies

QT Interval

QTc Corrected QT Interval

**QTcF** QT corrected with Fridericia's formula

RR Respiratory Rate
PT Preferred Term
RBC Red Blood Cell

SAE Serious Adverse EventSAP Statistical Analysis PlanSAS Statistical Analysis System

SD Standard Deviation
SOC System Organ Class

**SOPs** Standard Operation Procedures

**TEAEs** Treatment-Emergent Adverse Events

WBC White Blood Cell

WHO DD World Health Organization Drug Dictionary

mAbxience Research S.L.

#### 1. Introduction

This statistical analysis plan (SAP) is intended to give a detailed description of the summaries and the analyses that will be generated for the mAbxience Research S.L. study protocol No. MB02-A-06-20, Version 1.0, dated 26 May 2020 (Syneos Project No. 7012755). Safety and tolerability analyses will be described.

The plan may change due to unforeseen circumstances and any changes made after the plan has been finalized will be documented. If additional analyses are required to supplement the planned analyses described in the SAP, the changes and justification for the changes will be outlined in the Clinical Study Report (CSR). No change will be made without prior approval of the study Sponsor. No revision to the SAP is required for changes that do not affect the statistical analysis methods, definitions, or rules defined in this document.

When applicable, all methodology and related processes will be conducted according to Syneos's Standard Operating Procedures (SOPs) as appropriate. Protocol deviations occurring during the study will be listed.

Shells for all statistical tables, figures and listings referred to in this SAP will be displayed in a separate document. Statistical analysis plan and shells for PK analysis and immunogenicity analysis will be displayed in a separate document and it could be provided by Covance.



#### 2. Study Objectives

Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

#### 2.1 Primary objective

• To investigate and compare the pharmacokinetic (PK) profiles of MB02-SP (MB02 standard procedure), MB02-DM (MB02 defined media) and US-licenced Avastin® (US Avastin®) to establish bioequivalence between the 3 study arms.

#### 2.2 Secondary objectives

- Evaluation and comparison of derived PK parameters not covered by the primary endpoints for MB02-SP, MB02-DM and US Avastin®.
- To compare the safety profile of MB02-SP, MB02-DM and US Avastin<sup>®</sup>.
- To compare the immunogenicity of MB02-SP, MB02-DM and US Avastin<sup>®</sup>.



#### 3. Study Design

#### 3.1 General Design

This will be a Phase 1, double-blind, randomised, parallel-group, single-dose 3-arm study to investigate and compare the PK, safety and immunogenicity profiles of MB02-DM with MB02-SP and US Avastin® in healthy male subjects. A total of One hundred and fourteen (114) subjects will be randomised to one of following 3 arms in a 1:1:1 ratio:

- Arm 1: MB02-SP (MB02 standard procedure) as a 90 minute IV infusion
- Arm 2: MB02-DM (MB02 defined media) as a 90 minute IV infusion
- Arm 3: US Avastin® sourced from the US, as a 90 minute IV infusion.

Thirty-eight subjects will be dosed in each arm. Potential subjects will be screened to assess their eligibility to enter the trial within 30 days prior to study drug administration.

#### 3.2 Study Procedures

The overall schedule of procedures and assessments is provided in the protocol.

#### 3.3 Drug Administration

Subjects will receive a single dose of 1 mg/kg of one of the following treatments by IV infusion over 90 minutes. A total of 114 healthy adult male volunteers will be dosed; 38 subjects per treatment group, randomly assigned to one of the 3 treatment arms.

- 1 mg/kg dose of MB02-SP (bevacizumab biosimilar drug), administered as a 90 minute IV infusion.
- 1 mg/kg dose of MB02-DM (bevacizumab biosimilar drug), administered as a 90 minute IV infusion.
- 1 mg/kg dose of US Avastin<sup>®</sup>, administered as a 90 minute IV infusion.

#### 3.4 Subject Withdrawal and Replacement

A subject is free to withdraw from the study at any time. In addition, a subject will be withdrawn from dosing if any of the following criteria are met:

- Change in compliance with any inclusion/exclusion criterion that is clinically relevant and affects subject safety as determined by the Investigator (or designee);
- Noncompliance with the study restrictions that might affect subject safety or study assessments/objectives, as considered applicable by the Investigator (or designee);
- Any clinically relevant sign or symptom that in the opinion of the Investigator (or designee) warrants subject withdrawal.

mAbxience Research S.L.

If a subject is withdrawn from dosing, the Sponsor will be notified and the date and reason(s) for the withdrawal will be documented in the subject's electronic Case Report Form (eCRF). If a subject is withdrawn, efforts will be made to perform all Follow-up assessments, if possible. Other procedures may be performed at Investigator's (or designee's) and/or Sponsor's discretion. If the subject is in-house, these procedures should be performed before the subject is discharged from the clinic. The Investigator (or designee) may also request that the subject return for an additional Follow-up Visit. All withdrawn subjects will be followed until resolution of all their adverse events (AEs) or until the unresolved AEs are judged by the Investigator (or designee) to have stabilised.

Subjects who are withdrawn for nondrug related reasons may be replaced following discussion between the Investigator and the Sponsor. Subjects withdrawn as a result of AEs thought to be related to the study drug will generally not be replaced.

#### 3.5 Determination of Sample Size

Up to 114 subjects will be enrolled in order that 108 complete the study.

A sample size of 36 subjects per arm (108 subjects in total) will provide at least 90% power for all the pairwise comparisons for primary endpoints (AUC and Cmax) using a percent coefficient of variation (CV%) of 25% in both PK parameters for the similarity objective if the true ratio is equal to 1.05 or less.

A maximum of 5% loss of data due to premature discontinuation is expected therefore, the sample size is increased to 114 subjects in total, with 38 subjects per arm.

#### 3.6 Randomization and Blinding

A computer generated randomization schedule will be prepared by the assigned biostatistician prior to the start of the study. The schedule will be generated through the statistical analysis system (SAS) software, version 9.4. Subjects will be randomly assigned to 1 of 3 treatment arms and stratified into 2 groups based on weight ( $\geq$ 50.0 to <72.5kg, and  $\geq$ 72.5 to  $\leq$ 95.0 kg respectively).

For subjects who are replaced the replacements should take the same treatment assignment as the original subject to ensure that the planned treatment allocation ratio is retained.

The following controls will be employed to maintain the double blind status of the study:

• The Investigator and other members of staff involved with the study will remain blinded to the treatment randomisation code during the assembly procedure.

To maintain the blind, the Investigator will be provided with a sealed randomisation code for each subject, containing coded details of the treatment. These individual sealed envelopes will be kept in a limited access area that is accessible 24 hours a day. If, in order to manage subject safety (in the event of possibly treatment related SAEs or severe AEs), the decision to unblind resides with the Investigator. Whenever possible, and providing it does not interfere with or delay any decision in the best interest of the subject, the Investigator will discuss the intended code-break with the Sponsor. If it becomes necessary to break the code during the study, the date, time and reason will be recorded in the subject's source data and on the individual envelope and will be witnessed by a second person.



mAbxience Research S.L.

Where the subject experiences a suspected unexpected serious adverse reaction (SUSAR) the Sponsor pharmacovigilance team may be unblinded prior to notification of the relevant competent authorities and ethics committee in order to provide appropriate information.



#### 4. Changes from the Protocol

No changes in planned analyses were done compared to the protocol.



#### 5. Study Endpoints

#### 5.1 Primary Endpoints

The PK outcome endpoints of MB02-DM, MB02-SP and US Avastin® derived from the serum Concentration-time profile from Days 1 to 100 following IV administration are as follows:

- Area under the serum concentration-time curve from time zero to infinity  $(AUC_{[0-\infty]})$
- Maximum observed serum concentration (C<sub>max</sub>)

#### 5.2 Secondary Endpoints

- Evaluation of all other PK parameters for MB02-SP, MB02-DM and US Avastin<sup>®</sup>, including
  - $\circ$  Time of maximum observed serum concentration ( $t_{max}$ )
  - $\circ$  AUC from time zero to the time of the last observable concentration (AUC<sub>[0-t]</sub>)
  - o Clearance (CL)
  - $\circ$  Apparent serum terminal elimination half-life ( $t_{1/2}$ )
- The safety outcome measures for this study are as follows:
  - o Incidence and severity of AEs
  - Incidence of laboratory abnormalities, based on haematology, clinical chemistry, coagulation and urinalysis test results
  - o 12-lead electrocardiogram (ECG) parameters
  - Vital sign measurements
  - o Physical examinations

The immunogenicity of MB02-SP, MB02-DM and US Avastin®

 Determination of serum concentrations of anti-MB02-DM, MB02-SP, and anti-Avastin® antibodies.



#### 6. Analysis Populations

The analysis of safety and tolerability parameters will be based on the study population detailed in Section 6.1.

#### **6.1** Safety Population

The safety population will include all subjects exposed to MB02-DM, MB02-SP or US Avastin®, and have at least one post dose safety assessment.



#### 7. General Aspects for Statistical Analysis

#### 7.1 General Methods

SAS® for Windows, Release 9.4 (SAS® Institute Inc., Cary, NC, USA) software will be used to perform all data analyses.

All data in the database will be presented in the data listings. Unless otherwise stated, all listings will be sorted by randomized treatment group, subject number and assessment date/time

The following labels for treatment will be used on all tabulations where the results are displayed by treatment, in the following order:

- 1 mg/kg MB02 SP IV
- 1 mg/kg MB02 DM IV
- 1 mg/kg US Avastin® IV

#### 7.2 Summary Statistics:

Unless otherwise stated, continuous variables will be summarized using the number of observations (n), and the statistics mean, median, standard deviation (SD), minimum and maximum. The minimum and maximum values will be presented to the same number of decimal places as recorded in the case report form (CRF), mean and median will be presented to one more decimal place than the raw data and the SD will be presented to two more decimal places than the raw data. Summaries of change-from-baseline variables will include only subjects who have both a baseline value and corresponding value at the timepoint of interest. Categorical variables will be summarized with frequency counts and percentages. Percentages will be rounded to one decimal place, with the denominator being the number of subjects in the relevant population, unless otherwise stated.

Only data from nominal protocol scheduled visits will be included in the summary tables. Data from unscheduled visits will not be included in the summary tables (unless they were used as baseline) but will be included in the listings and figures.

#### 7.3 Key Definitions

Definition of Baseline

In general, base line will be defined for each subject and will be defined as the last available, non-missing assessment prior to first study drug administration. Unknown, Not Done, Not Applicable and other classifications of missing data will not be considered when calculating baseline observations. However, valid categorical observations will be considered for baseline calculations.

mAbxience Research S.L.

#### 7.4 Missing Data

All withdrawals will be included in all summaries up to the time of withdrawal.

There will be no imputation for missing data, unless otherwise specified.

#### 7.5 Visit Windows

All assessments will be included in the listings. No visit windows will be applied to assessments.

mAbxience Research S.L.

#### 8. Interim Analyses

No formal interim analysis was planned in the protocol.



#### 9. Study Population and Exposure

No inferential analysis will be done. Only observed data will be used.

#### 9.1 Subject Disposition

Subject disposition will be summarized by treatments (frequency and the percentage of subjects) and overall. The following categories will be summarized by number and/or percentage.

- Screened and screen failures subjects (overall only).
- Enrolled and not enrolled subjects (overall only).
- Subjects who are dosed in each treatment and overall.
- Subjects who have completed the study in each treatment and overall.
- Subjects who discontinued in each treatment and overall.
- Primary reason for discontinuation in each treatment and overall.

In addition, the number of randomized subjects, number of subjects evaluable for safety (Safety Population) will be presented by treatment and overall.

For subjects enrolled, not enrolled and screen failures, the percentage denominator will be the number of screened subjects. For all other calculations, the percentage denominator will be the number of subjects dosed in each treatment. For overall, the percentages will be based on the overall number of subjects dosed (safety population).

Subject study completion and discontinuation information will be listed. This listing will include the following information:

- Subject identifier and randomization number
- Study day/Date of informed consent
- Study day/Date of randomization (for randomized subjects)
- Study Treatment received (for randomized subjects)
- Study Day/ Date of study completion or discontinuation
- Primary reason for discontinuation

#### 9.2 Protocol Deviations

The protocol deviations will be categorized and listed by subject.

#### 9.3 Demographics and Baseline Characteristics

Descriptive statistics (sample size (n), mean, median, standard deviation [SD], minimum [Min], and maximum [Max]) will be calculated for continuous variables (age, body mass index [BMI],



mAbxience Research S.L.

height, and weight) considering last results (scheduled or unscheduled) obtained at screening. Frequency counts and percentages will be tabulated for categorical variables (gender, ethnicity, and race). All summaries will be presented by treatment for safety population. All demographic characteristics will be listed by subject.

#### 9.4 Medical History

Medical history will be listed by subject. The Medical Dictionary for Regulatory Activities (MedDRA®) Version 22.1 will be used to classify all medical history findings by System Organ Class (SOC) and Preferred Term (PT).

Urine drug screen, cotinine test and alcohol breath test will be listed only.

#### 9.5 Prior and Concomitant Medications

The use of prior and/or concomitant medications will be monitored throughout the study and listed by subject. The World Health Organization Drug Dictionary (WHO DD) Version Mar 2020, format B3 will be used to classify all medication reported during the study.

All prior and concomitant medications will be listed by subject.

#### 9.6 Study Drug Administration

The study drug administration details (including treatment received, infusion interruption, start and stop date and time of administration, total dose) will be listed by subject.



#### 10. Safety Analyses

Safety and tolerability data will be evaluated through the assessment of AEs, clinical laboratory parameters (clinical chemistry, hematology, cogulation, urinalysis and serology), 12-lead electrocardiogram (ECG), vital signs and physical examination. AEs, laboratory values, 12-lead ECG and vital signs will be summarized overall or according to the treatment, as appropriate. The analysis of the safety variables will be based on safety population.

Safety data will be summarized, but will not be subjected to inferential analysis.

#### **10.1** Physical Examination Findings

A full physical examination or symptom-directed physical examination will be performed at screening. Additionaly, symptom-directed physical examination will be performed at Day -1 (check-in) and Day 100 (End of Study (EOS)). A full physical examination or symptom-directed physical examination includes assessments of the following: Eye/Ear/Nose/Throat, General Appearance, Oral, Head and Neck, Chest/Lungs, Cardiovascular Abdomen, Musculoskeletal, Lymphatic, Dermatologic, Neurologic, Extremities, Psychiatric from the subject.

Body measurements, including height and body weight, will be measured and BMI will be calculated at screening. Body weight will also be measured at Day-1 (check-in). Body measurements will be summarized (mean, median, SD, min, max, and sample size) in demographic tables (safety population).

Any abnormal findings judged to be clinically significant will be documented as medical history or as an AE, during screening (non a TEAE) or after receiving treatment (TEAE). Any physical examination findings documented as AEs will be included in the AE summaries.

#### 10.2 Adverse Events

Treatment-emergent AEs (TEAEs) will be listed and summarised using descriptive methodology. TEAEs will be defined as AEs that occur on or after the date and time of study drug administration. Any AE that first occurs pre-dose but worsens in severity or is deemed to be related to the study drug after the first study drug administration will also be considered a TEAE. All AEs will be collected and documented during the course of the study. Subjects will be followed-up until final discharge from the study, and any AEs that occur during this time should be reported according to the procedures outlined below:

- All subjects with unresolved AEs at the end of the study, except those who dropped out before randomisation or starting active treatment, must be included in a safety follow-up visit to check response of AEs.
- Follow-up can be waived in specific cases after consultation with the Sponsor. This permission must be documented per case and retained in the Sponsor File.

The incidence of TEAEs and treatment-related AEs will be summarized using the safety population. The Medical Dictionary for Regulatory Activities (MedDRA®), Version 23.0 will be used to classify all AEs reported during the study by SOC and PT.



mAbxience Research S.L.

Incidence of subjects who experienced TEAEs (as well as number of events) will be presented by treatment and overall, by SOC, and PT, investigator-assessed relationship and also by severity. Each subject may only contribute once to each of the incidence rates, for a TEAE following a given treatment, regardless of the number of occurrences; the highest severity or highest relationship will be presented, as appropriate. In each table, SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

The causal relationship of an AE to the study drug will be assessed according to the study protocol as:

Not Related: when the AE is definitely caused by the subject's clinical state, or the

study procedure/conditions

Unlikely Related: when the temporal association between the AE and the drug is such that

the drug is not likely to have any reasonable association with the AE

Possibly Related: when the AE follows a reasonable temporal sequence from the time of

drug administration but could have been produced by the subject's clinical

state or the study procedures/conditions

Probably Related: when the AE has a reasonable time relationship to study drug

administration and is unlikely to be attributed to concurrent disease or

other drugs or chemicals

Related: when the AE follows a reasonable temporal sequence from administration

of the drug, abates upon discontinuation of the drug, follows a known or hypothesised cause-effect relationship, and (if appropriate) reappears when the drug is reintroduced. Treatment-related AEs will be those reported as Possibly Related, Probably Related or Related to Study Drug.

The severity of an AE or serious AE (SAE) will be recorded in the eCRF following the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, outlined below:

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only;

intervention not indicated

Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-

appropriate instrumental activities of daily living

Grade 3: Severe or medically significant but not immediately life-threatening;

hospitalisation or prolongation of hospitalisation indicated; disabling; limiting

self-care activities of daily living

mAbxience Research S.L.

Grade 4: Life-threatening consequences; urgent intervention indicated

Grade 5: Death related to AE

SAEs will be listed separately by subjects.

#### 10.3 Laboratory Parameters

Clinical laboratory (clinical chemistry, hematology, coagulation and urinalysis) results will be obtained at screening, Day -1 (check-in), Day 3, Day 8, Day 14, Day 21, Day 28, Day 42, Day 56, Day 78 and Day 100 (EOS).

Clinical chemistry parameters include the following: albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), Urea, low-density lipoprote in (LDL) cholesterol, high-density lipoprote in (HDL) cholesterol, triglycerides, total cholesterol, Uric acid, Calcium, Chloride, Inorganic phosphate, Potassium, Creatinine, Creatine kinase, Gamma-glutamyl transferase, Lactate dehydrogenase, Glucose, Sodium, Total bilirubin, Direct bilirubin, and Total protein.

Hematology parameters include the following: Haematocrit, Haemoglobin, Mean cell haemoglobin, Mean cell haemoglobin concentration, Mean cell volume, Platelet count, Red blood cell (RBC) count, White blood cell (WBC) count and WBC differentials as Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils.

Coagulation parameters include the following: International normalised ratio (INR), Prothrombin time and Activated partial thromboplastin time.

Urinalysis parameters include the following: Complete microscopic examination, pH, Specific gravity, Urobilinogen, Protein, Ketones, Blood, and Glucose. Unless otherwise specified, microscopic examination will be performed on abnormal findings and results will be listed.

Serology parameters including: Hepatitis B surface antigen (HBs Ag), Hepatitis B surface antibody (anti-HBs), Hepatitis B core antibody (anti-HBc), Hepatitis C antibody and Human immunodeficiency HIV antigen antibodies will be performed at screening.

Urinary drug screen including: Cotinine, Amphetamines/methamphetamines, Barbiturates, Benzodiazepines, Cocaine (metabolite), Methadone, Phencyclidine, Opiates, Tetrahydrocannabinoids, and Breath alcohol test will be performed at screening and at Day -1 (check-in).

Listings of all clinical laboratory results, including those unscheduled, will be provided with the abnormal values flagged with "L" for low and "H" for high for continuous parameters, and "A" for abnormal for categorical parameters.

Descriptive statistics (mean, median, SD, min, max, and sample size) for each clinical laboratory test (continuous variables) will be presented by treatment for each timepoints. Change from baseline descriptive statistics for post-dose measurements as well as for EOS will be presented. Baseline will be defined as the last results (scheduled or unscheduled) obtained prior to the study

mAbxience Research S.L.

drug administration. Unscheduled results will not be included in the summary tables except for baseline calculation if applicable. For categorical variables (urinalysis tests), the number of subjects (frequency and percentage) will be tabulated for each individual result (e.g., negative, positive, trace). Results from repeat tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an invalid initial result.

A summary table of shifts from baseline to EOS measurements will be provided. Baseline will be defined in the same manner as described in the preceding paragraph for continuous variables. The shift tables representing the categorical change of laboratory results (normal, abnormal not clinically significant, or abnormal clinically significant) from baseline to each post baseline visit will be presented. Results from repeat tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an invalid initial result.

If more than one clinical laboratory is used for the study, a formula that takes into consideration the relative normal ranges of each test of laboratories used will be applied to normalize these data. The conversion formula used will depend on the typical distribution of the normal range for each laboratory test; the two formula used are presented below:

 Hemoglobin, hematocrit, and platelet count test results are considered to have a normal distribution (Chuang-Stein, 1992) and the following formula will be used (Karvanen J., 2003):

$$S = L_s + (x-L_x) \frac{U_s-L_s}{U_x-L_x}$$

• The remaining hematology, biochemistry, and urinalysis test results are considered to have a non-normal distribution (Chuang-Stein, 1992) and the following formula will be used (Karvanen J., 2003):

$$s = \frac{x U_s}{U_x}$$

U= upper limit; L= lower limit; s= primary facility result; and x= secondary facility results.

Prior to applying these formulae, if required, units will be adjusted.

#### 10.4 Vital Signs

Supine blood pressure, supine pulse rate, respiratory rate (RR) will be assessed at screening, Day -1 (check-in), predose, 0.5H, 1H, End of infusion (EOI) and 2H of Day 1, Day 2, Day 5, Day 8, Day 10, Day 21, and Day 100 (EOS). Aural body temperature will be assessed at

mAbxience Research S.L.

screening, Day 2, Day 10, Day 21 and Day 100 (EOS) and pulse oximetry (PO) will be assessed at screening only.

Subjects must be supine for at least 5 minutes before blood pressure and pulse rate measurements.

Descriptive statistics (mean, median, SD, min, max, and sample size) will be presented by treatment for each timepoint and for each vital sign measurement. Change from baseline descriptive statistics for post-dose measurements as well as for EOS will be presented. Baseline will be defined as the last results (scheduled or unscheduled) obtained prior to the study drug administration. Unscheduled results will not be included in the summary tables except for baseline calculation if applicable. Results from repeat tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an invalid initial result.

A listing of all vital signs results will be provided by subject.

#### 10.5 Electrocardiogram

12-lead ECGs will be recorded after the subject has been supine and at rest for at least 5 minutes at screening, Day -1, Day 3, Day 8 and Day 100 (EOS). The quantitative ECG measurements are heart rate (HR), PR interval, QRS interval, QT interval, QTcF (Fridericia formula correction). Single 12 lead ECGs will be repeated once if either of the following criteria apply:

- QT interval corrected for heart rate using Fridericia's method (QTcF) > 500 msec
- QTcF change from the baseline (predose) is > 60 msec.

Descriptive statistics (mean, median, SD, min, max, and sample size) will be presented by treatment for each time point and for each ECG measurement. Change from baseline descriptive statistics for post-dose measurements as well as for EOS will be presented. Baseline will be defined as the last results (scheduled or unscheduled) obtained prior to the study drug administration. Unscheduled results will not be included in the summary tables except for baseline calculation if applicable. Results from repeat tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an invalid initial result.

Furthermore, a shift table representing the categorical change of ECGs results (normal, abnormal not clinically significant, or abnormal clinically significant) from baseline to each post baseline visit will be presented.

A listing of all ECG results will be provided with the abnormal values flagged.

Additionally, the listing of QT interval corrected for HR using Fridericia's method (QTcF) > 500 msec and QTcF change from the baseline (predose) is > 60 msec will be provided by subjects.

mAbxience Research S.L.

#### 11. Percentages and Decimal Places

If not otherwise specified, the following rules will be applied, with the exception of PK tables and listings described below:

- Percentages will be presented to one decimal place.
- Percentages equal to 0 or 100 will be presented as such without a decimal place.
- Minimum and maximum will be presented with the same precision as the original values;
   Mean, and median will be presented with one more decimal place than the original values, and standard deviation, will be presented with two more decimal place than the original values.



mAbxience Research S.L.

#### 12. Data Handling

The safety data will be received as SAS® datasets from the Syneos data management facility. Screening failures and ineligible volunteer's data (subject disposition) will be received from the clinical site as source data. The serum concentrations and Immunogenicity data will be provided by Covance.



#### 13. Handling of Missing Data

For safety,

- If an AE is recorded with an onset date corresponding to a dosing day, but the time is missing, then the AE will be assigned to the treatment.
- If an AE is recorded with an onset date that does not correspond to the dosing day, but the time is missing, then the AE will be assigned to the treatment if AE onset date is after dosing date.
- If an AE is recorded with an onset date where day and time are both missing, then the AE allocation to the treatment will be done on a case by case basis considering available information (e.g., AE onset date, AE end date, AE comments, subject disposition).

mAbxience Research S.L.

#### 14. Software to be Used

The safety data tables and listings will be created using SAS®, release 9.4. The study report text will be created using Microsoft® Office Word 2010, or a higher version.

mAbxience Research S.L.

#### 15. Reference List

- Chuang-Stein C. Summarizing laboratory data with different reference ranges in multicenter clinical trials. Drug Information Journal. 1992; 26:77-84.
- Karvanen J. The statistical basis of laboratory data normalization. Drug Information Journal. 2003; 37:101-107.

mAbxience Research S.L.

#### Table/Figure/Listing Shells (Without PK and Immunogenicity analysis)

A RANDOMISED, DOUBLE-BLIND, THREE-ARM, SINGLE DOSE, PARALLEL STUDY TO COMPARE THE PHARMACOKINETICS, SAFETY AND IMMUNOGENICITY OF MB02-SP, MB02-DM (BEVACIZUMAB BIOSIMILAR DRUGS) AND US LICENCED AVASTIN® IN HEALTHY MALE VOLUNTEERS

Sponsor Protocol No.: MB02-A-06-20 Syneos Health Clinique Inc. Project No.: 7012755

> Final Version: 1.0 Date: 26-MAY -2020

Contract Research Organization: Syneos Health, LLC/ Health UK Limited 1030 Sync Street, Morrisville, North Carolina 27560, United States Sponsor: mAbxience Research S.L. C/ Manuel Pombo Angulo, 28, 4<sup>th</sup> floor, 28050 Madrid, Spain

CONFIDENTIAL



mAbxience Research S.L.

## TABLE OF CONTENTS

| <b>TABL</b> | E OF CONTENTS | .32 |
|-------------|----------------------------------------------|------|
| 1. | Tables, Figures and Data Listings Formatting | .33 |
| | Table 1-1 Layout Specifications | .33 |
| 2. | Summary TFLs. | .34 |
| | Table 2-1 List of Table Shells | .34 |
| | Table 2-3 List of Data Listings Shells | .36 |
| 3. | CSR In-text Tables | .37 |
| 4. | Summary Tables | .40 |
| 5. | Listings | . 62 |

mAbxience Research S.L.

#### 1. Tables, Figures and Data Listings Formatting

The table, figure, and data listing (TFL) shells are presented in order to provide a framework for displaying the study data. The shells may change due to unforeseen circumstances. The shells may not be truly representative of every aspect of the study (e.g., sampling time points, assessed laboratory parameters, calculated parameters, units), but are intended to illustrate the general layout of the tables, figures, and data listings that will be included in the final report.

The default tables, listings, and figures layout will be as presented in Table 1-1:

**Table 1-1 Layout Specifications** 

| Orientation | Portrait | Landscape |
|-------------|---------------------------|-------------------|
| Paper Size | Letter | Letter |
| Margins | Top: 3.05 cm | Top: 3.05 cm |
| | Bottom: 2.54 cm | Bottom: 2.2 cm |
| | Left: 2.54 cm | Left: 1.9 cm |
| | Right: 2.54 cm | Right: 1.9 cm |
| Font | Table text: Times new Ro | oman 9 or 10 pts |
| | Table title: Times new Ro | oman 12 pts |
| | Table legend: Times new | Roman 9 or 10 pts |

The font size may be reduced as necessary to allow additional columns to be presented, but not at the expense of clarity. Also the orientation may be changed to portrait if appropriate.

#### 1.1 Headers

- All output should have the following header at the top left of each page:
- mAbxience Research S.L.
- All output should have Page n of N at the top or bottom right corner of each page. TLFs are internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where N is the total number of pages in the table).
- The date output was generated should appear along with the program name as a footer on each page.



# 2. Summary TFLs

## **Table 2-1 List of Table Shells**

| Table<br>Number | Title |
|---|---|
| | In-Text Table |
| 10.1-1 | Subject Disposition |
| | Demographic Data Summary Tables |
| 14.1-1 | Summary of Demographic Characteristics of Subjects Included in the Safety Population |
| 14.1-2 | Summary of Protocol Deviations – Safety Population |
| | Safety Data Summary Tables |
| 14.3.1-1 | Overview of Treatment-Emergent Adverse Events – Safety Population |
| 14.3.1-2 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events and Number of Events Summarized per Treatment – Safety Population |
| 14.3.1-3 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population |
| 14.3.1-4 | Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population |
| 14.3.1-5 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population |
| 14.3.1-6 | Number of Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population |
| 14.3.1-7 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Leading to Discontinuation Summarized per Treatment-Safety Population |
| 14.3.1-8 | Frequency of Subjects Experiencing Serious Treatment-Emergent Adverse Events Summarized per Treatment-Safety Population |
| 14.3.4-1 | Clinical Chemistry Summary Descriptive Statistics and Change from Baseline – Safety Population |
| 14.3.4-2 | Frequency of Subjects – Clinical chemistry Shifts from Baseline – Safety Population |
| 14.3.4-3 | Hematology Summary Descriptive Statistics and Change from Baseline – Safety Population |
| 14.3.4-4 | Frequency of Subjects – Hematology Shifts from Baseline – Safety Population |
| 14.3.4-5 | Urinalysis (pH and Specific Gravity) Summary Descriptive Statistics and Change from Baseline – Safety Population |
| 14.3.4-6 | Frequency of Subjects – Urinalysis (pH and Specific Gravity) Shifts from Baseline – Safety Population |
| 14.3.4-7 | Coagulation Summary Descriptive Statistics and Change from Baseline – Safety Population |
| 14.3.4-8 | Frequency of Subjects - Coagulation Shifts from Baseline - Safety Population |
| 14.3.4-9 | Urinalysis Frequency Summary – Categorical Results – Safety Population |
| 14.3.4-10 | Frequency of Subjects – Urinalysis Shifts from Baseline – Categorical Results – Safety Population |
| 14.3.4-11 | Vital Signs Summary Descriptive Statistics and Change from Baseline – Safety Population |
| 14.3.4-12 | Electrocardiograms Summary Descriptive Statistics and Change from Baseline – Safety Population |



mAbxience Research S.L.

| 14.3.4-13 | Frequency of Subjects – Electrocardiograms Shifts from Baseline – Safety Population |
|---|---|


mAbxience Research S.L.

### Table 2-3 List of Data Listings Shells

| Listing<br>Number | Title |
|---|---|
| | Subject Characteristics Listings |
| 16.2.1-1 | Subjects Completion and Discontinuation Information |
| 16.2.2-1 | Protocol Deviations Protocol Deviations |
| 16.2.4-1 | Demographics |
| 16.2.4-2 | Medical History Findings at Screening |
| 16.2.4-3 | Prior and Concomitant Medications |
| 16.2.4-4 | Study Drug Administration |
| 16.2.4-5 | Interruption of IV Infusion |
| 16.2.4-6 | Assignments to Analysis Populations |
| 16.2.4-7 | Cotinine Test |
| 16.2.4-8 | Urine Drug Screen |
| 16.2.4-9 | Alcohol Breath Test |
| 16.2.4-10 | Randomization |
| | Safety Data Listings |
| 16.2.7-1 | Non-Treatment-Emergent Adverse Events |
| 16.2.7-2 | Treatment-Emergent Adverse Events |
| 16.2.7-3 | Serious Adverse Events |
| 16.2.7-4 | Treatment-Emergent Adverse Events with NCI-CTCAE of Grade 3 or Higher |
| 16.2.7-5 | Treatment-Emergent Adverse Events Leading to Study Drug Withdrawal/Discontinuation |
| 16.2.8-1 | Clinical Laboratory – Clinical chemistry |
| 16.2.8-2 | Clinical Laboratory – Hematology |
| 16.2.8-3 | Clinical Laboratory – Urinalysis |
| 16.2.8-4 | Clinical Laboratory – Coagulation |
| 16.2.8-5 | Clinical Laboratory – Serology |
| 16.2.8-6 | Clinical Laboratory – Urine Drug Screen and Alcohol Breath Tests |
| 16.2.8-7 | Vital Signs Result |
| 16.2.8-8 | Pulse oximetry Results |
| 16.2.8-9 | ElectrocardiogramResult |
| 16.2.8-10 | QT interval corrected for heart rate using QTcF > 500 ms ec |
| 16.2.8-11 | QTcF change from the baseline (predose) is > 60 msec |
| 16.2.8-12 | Physical Examination Findings by Subject |



mAbxience Research S.L.

### 3. CSR In-text Tables



mAbxience Research S.L.

| Category | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | 1 mg/kg US - Avastin® IV | Overall |
|---|---|---|---|---|
| Screened | | | | xx |
| Screening Failures <sup>1,2</sup> | | | 1 | x ( xx.x) |
| Not Enrolled <sup>1,3</sup> | | | 1 | x ( xx.x) |
| Enrolled <sup>1,4</sup> | | 1 | 1 | x ( xx.x) |
| Safety Population | x ( xx.x) | x ( xx.x) | x (xx x) | x (xx.x) |
| Randomized | XX | XX | XX | xx |
| Dosed | XX | XX | XX | XX |
| Not Dosed | XX | XX | XX | XX |
| Completed Study <sup>5,6</sup> | x (xx.x) | x ( xx.x) | x ( xx x) | x ( xx.x) |
| Number of Subjects Discontinued <sup>7</sup> | XX | XX | XX | XX |
| Primary Reason for Discontinuation 7,8 | | | | |
| Adverse Event | x ( xx.x) | x ( xx.x) | x (xx x) | ( x.x.x) |
| Death | x ( xx.x) | x ( xx.x) | x (xx x) | x(xx.x) |
| Lost To Follow-up | x (xx.x) | x (xx.x) | x ( xx x) | (x.x.x) |
| Physician Decision | x ( xx.x) | x ( xx.x) | x ( xx x) | (x.x.x) |
| ProtocolDeviation | x ( xx.x) | x ( xx.x) | x ( xx x) | ( xx.x) |
| Study Terminated by Sponsor | x ( xx.x) | x ( xx.x) | x ( xx x) | x ( xx.x) |
| InformedConsent Withdrawn | x ( xx.x) | x ( xx.x) | x ( xx x) | (xx.x) |
| Withdrawal by Subject | x ( xx.x) | x (xx.x) | x (xx x) | x (xx.x) |
| Other | ( ^ ^ ^ ) ^ | (^ ^^ ) ^ | (^ ^^ ) ^ | ( ^ ^ ) ^ |

Percentage based on the number of screened subjects.

<sup>2</sup> Screening failures include subjects who did not meet project criteria.

<sup>3</sup> Not enrolled include subjects who were judged eligible but decided not to participate on study or who were not selected to participate in the study since there was already a sufficient number of subjects.



mAbxience Research S.L.

<sup>4</sup> Enrolled include subjects who were judged eligible and accepted to participate in the trial after having signed the approved final version of the study informed consent form and also those identified as standby who may replace subjects who withdraw from the study before dosing.

<sup>5</sup> Completed study include subjects who complete the study until follow-up visit without major protocol deviation.

<sup>6</sup> Percentage based on the number of dosed subjects for a given treatment.

7 Overall, each subject could only contribute once to each reason for discontinuation, regardless of the number of occurrences.

<sup>8</sup> Percentage based on the number of discontinued subjects per treatment group or overall, as appropriate.

Data source: Listings 16.2.1-1 and 16.2.4-4.

20 May 2021 (Final 1.0)



mAbxience Research S.L.

### 4. Summary Tables



mAbxience Research S.L.

| Category | Statistic | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | $1 \mathrm{mg/kg} \mathrm{US}$ - $\mathrm{Avastin}^{\circledast} \mathrm{IV}$ |
|---|---|---|---|---|
| Age (years) | Z | xx | xx | XX |
| | Mean | x xx | XX.X | X XX |
| | SD | x xx | XX.X | X XX |
| | Median | x xx | XX.X | X XX |
| | Min, Max | XX-XX | XX-XX | XX-XX |
| Gender | | | | |
| Male | n (%) | x (xxx) | ( x x x ) x | x ( xx.x) |
| Ethnicity | | | | |
| Not Hispanic or Latino | n (%) | x (xx x) | x ( xx x) | x (xx.x) |
| Hispanic or Latino | n (%) | x (xxx) | x (xx x) | x (xx.x) |
| Not Reported | n (%) | x (xx x) | x ( xx x) | x (xx.x) |
| Unknown | n (%) | x (xxx) | x (xx x) | x (xx.x) |
| Asian | (%) " | ( ^ | ( ^ ^ ^ | ( ^ ^ ^ ) ^ ^ |
| Asian | n (%) | ( | ( | x ( xx.x ) |
| Black | n (%) | x (xxx) | X(XXX) | X(XX.X) |
| Australian Aborigine/Torres Strait Islander | n (%) | x (xxx) | x ( xx x) | x (xx.x) |
| Pacific Islander | n (%) | x (xxx) | x ( xx x) | x ( xx.x) |
| White | n (%) | x (xxx) | x (xx x) | x (xx.x) |
| Other | n (%) | x (xxx) | x (xx x) | x ( xx.x) |
| Height (cm) | Z | XX | XX | XX |
| | Mean | XX.XX | XX XX | XX.XX |
| | SD | XX.XX | XX XX | XX.XX |
| | Median | XX.XX | XX XX | XX.XX |
| | Min, Max | XX XX-XX XX | XX.XX-XX.XX | XX XX-XX XX |
| Weight (kg) &reening | z | XX | XX | XX |
| | Mean | XX.XX | XX XX | XX.XX |
| | 9 | | | |


20 May 2021 (Final 1.0)



mAbxience Research S.L.

| | Median<br>Min, Max | XX.XX<br>XX XX-XX XX | XX XX<br>XX.XX-XX.XX | XX.XX<br>XXXX-XX XX |
|---|---|---|---|---|
| Weight (kg) Day -1 | N<br>Mean<br>SD<br>Median<br>Min, Max | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX XX<br>XX XX<br>XX XX<br>XX XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX |
| Weight (≥50.0 to <72.5 kg) (kg) | N<br>Mean<br>SD<br>Median<br>Min, Max | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX XX<br>XX XX<br>XX XX<br>XX XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX |
| Weight (≥72.5 to ≤95.0 kg) (kg) | N<br>Mean<br>SD<br>Median<br>Min, Max | XX XX.XX XX X | XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX |
| $ m BMI(kg/m^2)$ | N<br>Mean<br>SD<br>Median<br>Min, Max | XX XXX<br>XX XXX<br>XX XXX<br>XX XXX XX | XX XXX XX XXX XX XXX XX XXX XX XXX | XX<br>XX XXX<br>XX XXX<br>XX XXX XX |

Programming Note: 1) Refer to the note below for additional instructions

N: Number of subjects dosed; n (%): Number and percent of subjects; SD: Standard Deviation. Am Indian: American Indian or Alaskan Native; Black: Black or African American;

BMI: body mass index.



mAbxience Research S.L.

Last results (scheduled or unscheduled) obtained at screening were used to generate this table. Data source: Listing 16.2.4-1


20 May 2021 (Final 1.0)



mAbxience Research S.L.

# Table 14.1-2 Summary of Protocol Deviations - Safety Population

| Protocol Deviation Category | 1 mg/kg MB02 - SP IV $(N=xxx)$ | 1 mg/kg MB02 - DM IV<br>(N= xxx) | 1 mg/kg US - Avastin <sup>®</sup> IV<br>(N= xxx) |
|---|---|---|---|
| | | | ; |
| Category 1 | XX (XX.X%) | xx (xx.x%) | xx (xx.x⋄) |
| Category 2 | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) |
| Category 3 | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) |
| etc | (×.xx) xx | xx (xx.x%) | xx (xx.x%) |

Programming Notes: Include categories as available in the source protocol deviation log.



mAbxience Research S.L.

| Table 14.3.1-1 Overview of Treatment-Emergent Adverse Events – Safety Population | atment-Eme | rgent Adverse Event | s – Safe ty Population | | |
|---|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA® Preferred Term | Statistic | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | 1 mg/kg US - Avastin® IV | Overall $(N=XX)$ |
| Subjects with TEAEs | (%) u | ( x.x. ) x | x (xx x) | x (xx.x) | x (xx x) |
| Number of TEAEs | [E] | [x] | [x] | [x] | [x] |
| Subjects with SAEs | n(%) | x (xx.x) | x (xx x) | x (xx.x) | x (xxx) |
| Total number of SAEs | [E] | [x] | [x] | [x] | [x] |
| Subjects discontinued due to TEAEs | n(%) | x (xx.x) | x ( xx x) | x(xx.x) | x (xx x) |
| Total number of TEAEs leading to discontinuation | [E] | [x] | [x] | × | [x] |
| All TEAEs by Severity Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life Threatening Grade 5: Death Total | n(%)[E]<br>n(%)[E]<br>n(%)[E]<br>n(%)[E]<br>n(%)[E] | [x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x | x (xxx) x<br>x (xxx) x<br>x (xxx) x<br>x (xxx) x<br>x (xxx) x<br>x (xxx) x<br>x (xxx) x | x ( xx x ) x | x (xx x) [x]<br>x (xx x) [x]<br>x (xx x) [x]<br>x (xx x) x<br>[x] (x xx ) x<br>[x] (x xx x) x |
| Related TEAEs (possible, probable, related) by severity Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life Threatening Grade 5: Death Total | n (%)[E]<br>n (%)[E]<br>n (%)[E]<br>n (%)[E]<br>n (%)[E] | [x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x | x (xxx x) x | x (xx x) x<br>x (xx x) x<br>[x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x | [x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x<br>[x] (x xx ) x |

E: Number of TEAEs; N: Number of subjects dosed; n (%): Number and percent of subjects with TEAE; MedDRA ®: Medical Dictionary for Regulatory Activities, version 23.0; TEAEs: Treatment-Emergent Adverse Events.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences. Overall: Included results from all treatment groups.



mAbxience Research S.L.

Table 14.3.1-2 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events and Number of Events Summarized per Treatment - Safety Population

| Tradilicit — Saicty Topulation | ILUII | | | | |
|---|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA® Preferred Term | Statistic | 1 mg/kg MB02 - SP IV<br>(N=XX) | 1 mg/kg MB02 - DM IV<br>(N=XX) | 1 mg/kg US - Avastin® IV<br>(N=XX) | Overall (N=XX) |
| Number of TEAEs<br>Number of Subjects with TEAEs | E<br>n (%) | xx<br>x (xx.x) | xx<br>x (xx x) | xx<br>x (xx.x) | xx x (xx x) |
| MedDRA® System Organ Class 1<br>MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | n(%) [E]<br>n(%) [E]<br>n(%) [E] | x (xxx) x<br>[x] (xxx) x<br>[x] (xxx) x | x (xx.x)[x]<br>x (xx.x)[x]<br>x (xx.x)[x] | $\begin{array}{c} x (xxx)[x] \\ x (xxx)[x] \\ x (xxx)x \end{array}$ | x (xx x) [x] x (xx x) x [x] (x xx ) x [x] (x xx ) x |
| MedDRA® System Organ Class 2<br>MedDRA® Preferred T erm 1<br>MedDRA® Preferred T erm 2 | n(%) [E]<br>n(%) [E]<br>n(%) [E] | $\begin{array}{c} x(xxx)x\\ x(xxx)x\\ x(xxx)x \end{array}$ | x (xx.x) [x]<br>x (xx.x) [x]<br>x (xx.x) [x] | x(xxx)[x] $x(xxx)[x]$ $x(xxx)[x]$ | $\begin{array}{c} x(xxx)[x] \\ x(xx)x \\ x(xx)[x] \end{array}$ |
| MedDRA® System Organ Class 3<br>MedDRA® Preferred T erm 1<br>MedDRA® Preferred T erm 2 | n(%) [E]<br>n(%) [E]<br>n(%) [E] | $\begin{array}{c} x(xxx)x\\ x(xxx)x\\ x(xxx)x \end{array}$ | x (xx.x) [x]<br>x (xx.x) [x]<br>x (xx.x) [x] | x(xxx)[x] $x(xxx)[x]$ $x(xxx)[x]$ | $ \begin{array}{c} x(xxx)[x] \\ x(xx)[x] \\ x(xx)[x] \end{array} $ |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

2) Refer to footnotes for additional instructions.

E: Number of TEAEs; N: Number of subjects dosed; n (%): Number and percent of subjects with TEAE; MedDRA ®: Medical Dictionary for Regulatory Activities, version 23.0; TEAEs: Treatment-Emergent Adverse Events.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences.

Overall: Included results from all treatment groups.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analys is Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

Table 14.3.1-3 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class | | | 1 mg/kg MB02 - SP IV | 02 - SP IV | | | | | 1 mg/kg N | 1 mg/kg MB02 - DM IV | VI | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® PreferredTerm | | | <u>(</u> ) | (N=XX) | | | | | J) | (N=XX) | | |
| n (%) | n (%) Grade 1 Grade 2 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 3 Grade 4 Grade 5 TotalTEAEs | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 1 Grade 2 Grade 3 Grade 4 Grade 5 Total TEAEs |
| MedDRA® System Organ Class 1 | x (xx.x) | x(xx.x) x(xx.x) | (x xx) | x(xxx) | (x xx) | x ( xx x) | x ( xx x) | (x.x.) | $(x \times x)$ | x(xxx) $x(xxx)$ $x(xxx)$ | (x.x.) | (xx.x) |
| MedDRA® Preferred Term 1 | x(xx.x) | (x.x.x) | $(x \times x)$ | $(x \times x)$ | $(x \times x)$ | $(x \times x)$ | x(xxx) | x(xx.x) | $(x \times x)$ | $(x \times x)$ | x(xx.x) | (xx.x) |
| MedDRA® Preferred Term 2 | x(xx.x) | (x.x.x) | (x xx) | (x xx) | (x xx) | x ( xx x) | (x xx) | x(xx.x) | (x xx) | (x xx) | (x.x.x) | (x.x.x) |
| MedDRA® System Organ Class 2 | x (xx.x) | x(xx.x) x(xx.x) | $(x \times x)$ | $(x \times x)$ | $(x \times x)$ | ( x x x ) x | x ( xx x) | x(xx.x) | x(xxx) | (xx x) x (xx x) | x(xx.x) | x(xx.x) |
| MedDRA® Preferred Term 1 | x (xx.x) | (x.x.x) | $(x \times x)$ | $(x \times x)$ | $(x \times x)$ | $(x \times x)$ | x(xxx) | x(xx.x) | $(x \times x)$ | $(x \times x)$ | x(xx.x) | (xx.x) |
| MedDRA® Preferred Term 2 | x (xx.x) | x(xx.x) | (x xx) | (x xx) | (x xx) | x ( xx x) | (x xx)x | (xx.x) | (x xx) | (x xx) | (x.x.x) | x(xx.x) |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equalrates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity. 3)

Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse events; MedDRA ®: Medical Dictionary for Regulatory Activities, version 23.0.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest severity is presented.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3: Severe or medically significant but not immediately life-threatening; hos pitalis ation or prolongation of hospitalisation indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.

Fotal TEAEs: Includes results from all severities per treatment and overall.

Overall: Included results from all treatment groups.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analys is Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

Table 14.3.1-3 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Ponulation (cont.)

| Saicty robulation (cont.) | [-] | | | ( | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | | 1 mg/kg US<br>(N | 1 mg/kg US - Avastin®IV<br>(N=XX) | ΛI | | | | Overall<br>(N=XX) | rall<br>XX) | | |
| n (%) | | Grade 1 Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 4 Grade 5 Total TEAEs Grade 1 | Grade 1 | Grade 2 | Grade 3 | Grade 3 Grade 4 | Grade 5 | Total<br>TEAEs |
| MedDRA® System Organ Class x (xx x) x (xx.x) | x ( xx x) | x (xx.x) | x ( xx.x) | xx.x) x (xx.x) x (xx x) | ( x x x ) x | ( x x x ) x | x (xx.x) | x (xx.x) x (xx x) | x (xx.x) | x (xxx) x (xxx) x (xxx) | x (xx x) | x (xxx) |
| MedDRA® PreferredTerm 1<br>MedDRA® PreferredTerm 2 | x (xx x)<br>x (xx x) | x(xx x) x(xx.x)<br>x(xx x) x(xx.x) | x (xx.x)<br>x (xx.x) | x (xx.x)<br>x (xx.x) | x ( xx x)<br>x ( xx x) | x ( xx x)<br>x ( xx x) | x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x) | x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x) | x ( xx x)<br>x ( xx x) | x (xx x)<br>x (xx x) |
| MedDRA® System Organ Class $x(xx x) x(xx x)$ | x (xx x) | x (xx.x) | x (xx.x) | X(XX.X) X(XX.X) | (x xx) | x (xx x) | x (xx.x) | ( x x x ) | x (xx.x) | x (xxx) | x (xx x) | x (xxx) |
| Z<br>MedDRA® PreferredTerm 1<br>MedDRA® PreferredTerm 2 | x ( xx x ) x x ( x x x ) x | x ( xx x) x ( xx.x) x ( xx.x) x ( xx x) x ( xx.x) | x (xx.x)<br>x (xx.x) | x (xx.x)<br>x (xx.x) | x ( xx x)<br>x ( xx x) | x ( xx x)<br>x ( xx x) | x (xx.x)<br>x (xx.x) | x (xx x)<br>x (xx x) | x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x) | x (xx x)<br>x (xx x) | x (xx x)<br>x (xx x) |

Programming Notes:

SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity 35

Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse events; MedDRA ®: Medical Dictionary for Regulatory Activities,

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalisation of hospitalisation indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest severity is presented. intervention indicated; Grade 5: Death related to AE.

Total TEAEs: Includes results from all severities per treatment and overall.

Overall: Included results from all treatment groups.



mAbxience Research S.L.

| Table 14.3.1-4 Number of Treatment-Emergent | atment- | Emerge | nt Adve | Adverse Even | nts Sumn | narized per Trea | Treatme | ent and § | Severity | t and Severity – Safety | y Popula | tion |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | | /kg M | B02 - SP IV<br>N=XX) | , | | | | 1 mg/kg MB02<br>(N=XX | MB02 - DM<br>(N=XX) | 1 IV | |
| I | E Grade 1 Grade 2 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | TotalTEAEs | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Total TEAEs |
| Total Number of TEAEs | | | | | | | | | | | | |
| MedDRA® System Organ Class 1 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® PreferredTerm 1 | × | × | × | × | × | X | × | × | × | × | × | × |
| MedDRA® Preferred Term 2 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® System Organ Class 2 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® PreferredTerm 1 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® Preferred T erm 2 | × | × | × | × | × | × | × | × | × | × | × | × |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equalrates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3: Severe or medically significant but not immediately life-threatening; hos pitalisation or prolongation of hospitalisation indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 23.0. intervention indicated; Grade 5: Death related to AE.

Total TEAEs: Includes results from all severities per treatment and overall.

Overall: Included results from all treatment groups.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analys is Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

| Table 14.3.1-4 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population (cont | rofTrea | tment-En | nergent A | dverse E | vents Sumr | narized pe | er Treatm | ent and S | everity – | Safe ty Pop | oulation ( | cont.) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® System Organ<br>Class<br>MedDRA® PreferredTerm | | | 1 mg/kg US | US - Avastin® IV<br>(N=XX) | > | | | | O <sub>v</sub> | Overall (N=XX) | | |
| Ξ | | Grade 1 Grade 2 Grade 3 | Grade 3 | Grade 4 | Grade 5 | Total<br>TEAEs | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Total<br>TEAEs |
| Total Number of TEAEs ModDDA® System Organ | > | > | > | > | > | > | > | > | > | > | > | > |
| Class 1 MedDRA® Preferred Term 1 | < × | < × | < × | < × | < × | < × | < × | < × | < × | < × | < × | < × |
| MedDRA <sup>®</sup> PreferredTerm 2 | : × | × | · × | : × | : × | · × | : × | × | : × | × | × | : × |
| MedDRA® System Organ | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® PreferredTerm 1 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® Preferred Term 2 | × | × | × | × | × | × | × | × | × | × | × | × |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity. 35

Refer to footnotes for additional instructions.

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting self-care activities of daily living; Grade 4: Life-threatening consequences; urgent E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA ®: Medical Dictionary for Regulatory Activities, version 22.1 intervention indicated; Grade 5: Death related to AE.

Total TEAEs: Includes results from all severities per treatment and overall.

Overall: Included results from all treatment groups.



mAbxience Research S.L.

# Table 14.3.1-5 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship - Safety Population

| MedDRA® System Organ | | | 1 mg/k | 1 mg/kg MB02 - SP IV | VI q | | | | 1 mg/ | 1 mg/kg MB02 - DM IV | DM IV | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class<br>MedDRA® Preferred Term | | | | (N=XX) | | | | | | (N=XX) | | |
| (%) u | Not | Not Unlikely Possibly | Possibly | Probably | Probably Related | Total related TEAEs | Not | Unlikely | Possibly | Probably | Related | Unlikely Possibly Probably Related Total related TEAEs |
| | related | related related | related | related | | $ \begin{array}{c c} (possibly + probably + \\ \hline related & related \\ \hline \end{array} $ | related | related | related | related | | (possibly + probably + related) |
| ModDD A ® Syntam Owns | (3, 3,3, ) | (,, ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | (* **, | (" "") " | (", ",") ", | | , (,, ,,,, ) | (", "", | (* ***) ** | (* ***) ** | (" "") " | (" "") " |
| Class 1 | ( v.v.v ) v | ( | (x.xx.) x | ( | ( v.v. ) v | ( | ( (v vv ) v | ( | ( | ( | ( y.y.y ) y | ( v. v. v ) v |
| MedDRA® PreferredTerm 1 x (xx.x) x (xx x) x (xx.x) | x (xx.x) | (x xx) x | x (xx.x) | (x.xx)x(xx.x) | x (xx.x) | x (xxx) | x (x xx) x | ( x x x ) | ( x x x ) x | x(xx) x(xxx) x(xxx) x(xxx) | x (xx.x) | x (xx.x) |
| MedDRA® Preferred Term 2 x (xx.x) x (xx x) x (xx.x) | x (xx.x) | ( x x x ) x | x (xx.x) | (x.xx)x(xx.x)x | x (xx.x) | x (xxx) | x (x xx) x | ( | x(xxx)x(xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | , | , | , | , | | , | , | , | , | , | , |
| MedDRA® System Organ | x ( xx.x) | x ( xx.x) x ( xx x) x ( xx.x) | x ( xx.x) | x (xx x) x (xx.x) | x (xx.x) | x (xxx) | x (xx x) x | ( xx x) | ( x x x ) x | x(xx)x(xx) $x(xx)$ $x(xx)$ | x ( xx.x) | x ( xx.x) |
| MedDRA® PreferredTerm 1 x (xx.x) x (xx x) x (xx.x) | x (xx.x) | x ( xx x) | x (xx.x) | $(x \times x) \times (x \times x)$ | x (xx.x) | x (xx x) | x (x xx) x | (x xx ) | x ( x x x ) x ( x x x ) x ( x x x ) x ( x x x ) | x (xx.x) | x ( xx.x) | x (xx.x) |
| $MedDRA^{\circledast} \ PreferredTerm \ 2 \ \ x \ (xx.x) \ \ x \ (xx.x) \ \ x \ (xx.x)$ | x (xx.x) | (x xx) | x(xx.x) | x(xxx) x(xxx) | x(xx.x) | x (xxx) | x (x xx) x | ( x x x ) | x(xxx) x(xxx) x(xxx) x(xxx) | x(xx.x) | x(xx.x) | x (xx.x) |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equalrates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.

3) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse event; MedDRA ®: Medical Dictionary for Regulatory Activities, Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences; the highest relationship is presented. version 23.0

Total related TEAEs: Includes results from possibly, probably and related relationships per treatment and overall.

Overall: Included results from all treatment groups.



mAbxience Research S.L.

# Table 14.3.1-5 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationshin - Safety Pounlation

| relations in parety i option | I Opula | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® System Organ<br>Class<br>MedDRA® Preferred Term | | | l mg/kg | kg US - Ava | US - Avastin <sup>®</sup> IV<br>(N=XX) | | | | | Overall<br>(N=XX) | | |
| n (%) | Not<br>related | Not Unlikely Possibly<br>related related related | Possibly<br>related | Probably<br>related | Related | Probably Related TotalrelatedTEAEs Not Unlikely related (possibly + probably + related related related) | | Jnlikely<br>related | Possibly<br>related | Probably<br>related | Related | Related Total related TEAEs<br>(possibly + probably + related) |
| MedDRA® System Organ<br>Class 1 | x (xxxx) | x ( xx x) | x (xxx) x (xx x) x (xx.x) | x (xxx) x (xxx) | x (xx.x) | ( x x x ) x | x (x xx) x | (x xx ) | x (xx x) | x(xx) x (xxx) x (xxx) x (xxx) x | x ( xx.x) | x (xx.x) |
| $MedDRA^{\circledast} \ Preferred Term \ 1 \ \ x \ x.x.x) \ x \ (xx.x) \ x \ (xx.x)$ | x (xx.x) | (x xx) x | (x.x.) | x(xxx) x(xxx) | x (xx.x) | $(x \times x)$ | x (x xx) x | (x xx) | ( x x x ) x | x(xx x) x(xx x) x(xx x) x(xx x) | x(xx.x) | x (xx.x) |
| MedDRA <sup>®</sup> Preferred Term 2 x (xx.x) x (xx x) | x ( xx.x) | x (xx x) | x (xx.x) | x (xx x) x (xx.x) | x (xx.x) | x (xx x) | x (x xx) x | (x xx ): | x (xxx) x (xxx) x (xxx) | x ( xx.x) | x (xx.x) | x (xx.x) |
| MedDRA® System Organ<br>Class 2 | x ( xx.x) | x (xx.x) x (xx x) x (xx.x) | x (xx.x) | x (xx x) x (xx.x) | x (xx.x) | x (xxx) | x (x xx) x | ( xx x) | x (x xx ) | (xx x) x (xx x) x (xx x) x (xx x) x (xx xx) | x (xx.x) | x (xx.x) |
| $\label{eq:medDRA} MedDRA^{\circledast} \ PreferredTerm \ 1 \ x(\ xx.x) \ x(\ xx.x) \ x(\ xx.x) \\ MedDRA^{\circledast} \ PreferredTerm \ 2 \ x(\ xx.x) \ x(\ xx.x) \ x(\ xx.x) \\$ | x ( xx.x)<br>x ( xx.x) | x ( xx x)<br>x ( xx x) | x (xx.x)<br>x (xx.x) | x (xx x) x (xx.x)<br>x (xx x) x (xx.x) | x (xx.x)<br>x (xx.x) | x (xx x)<br>x (xx x) | x (x xx) x x (x xx) x | (x xx ): | x ( xx x)<br>x ( xx x) | x (xx x) x (xx x) x (xx x) x (xx.x) | x ( xx.x)<br>x ( xx.x) | x (xx.x)<br>x (xx.x) |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equalrates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.

() Refer to footnotes for additional instructions.



mAbxience Research S.L.

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | | 1 mg/k | 1 mg/kg MB02 - SP IV<br>(N=XX) | SP IV | | | | 1 mg/ | 1 mg/kg MB02 - DM IV<br>(N=XX) | DM IV | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| B | Not<br>related | Not Unlikely Possibly<br>related related related | Possibly related | Probably Related<br>related | | Total related TEAEs<br>(possibly + probably + related) | Not<br>related | Unlikely<br>related | Possibly related | Probably<br>related | Related | Probably Related Total related TEAEs related (possibly + probably + related) |
| MedDRA® System Organ Class | × | × | × | × | × | × | × | × | × | × | × | X |
| MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | × × | × × | × × | × × | × × | × × | × × | × × | × × | × × | × × | × × |
| MedDRA® System Organ Class<br>2 | × | × | × | × | × | × | × | × | × | × | × | × |
| $MedDRA^{\otimes}$ Preferred Term 1 | × | × | × | × | × | × | × | × | × | × | × | × |
| $MedDRA^{\circledast}$ Preferred Term 2 | × | × | × | × | × | × | × | × | × | × | × | × |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equalrates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 23.0 Total related TEAEs: Includes results from possibly, probably and related relationships per treatment and overall. Overall: Included results from all treatment groups. Data source: Listing 16.2.7-2



mAbxience Research S.L.

| MedDRA® System<br>Organ Class<br>MedDRA®<br>Preferred Term | | | 1 mg/kg U | 1 mg/kg US - Avastin <sup>®</sup> IV<br>(N=XX) | >. | | | | <b>3</b> () | Overall (N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | E Not related Unlikely related | Unlikely<br>related | Possibly related | Probably<br>related | Related | Total related<br>TEAEs (possibly<br>+ probably +<br>related) | Not<br>related | Unlikely<br>related | Possibly related | Probably<br>related | Related | Total related<br>TEAEs (possibly<br>+ probably +<br>related) |
| MedDRA® System | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® PreferredTerm 2 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® System | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® Dreferred Term 1 | × | × | × | × | × | × | × | × | × | × | × | × |
| MedDRA® PreferredTerm 2 | × | × | × | × | × | × | × | × | × | × | × | × |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship 7

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 22.1. Total related TEA Es: Includes results from possibly, probably and relate drelationships per treatment and overall. Overall: Included results from all treatment groups.



mAbxience Research S.L.

Table 14.3.1-7 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Leading to Discontinuation Summarized per Treatment - Safety Population

| per ricaminant – Saiciy ropulation | папоп | | | | |
|---|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA® Preferred Term | Statistic | 1 mg/kg MB02 - SP IV<br>(N=XX) | 1 mg/kg MB02 - DM IV<br>(N=XX) | 1 mg/kg US - Avastin® IV<br>(N=XX) | Overall (N=XX) |
| Number of Subjects with TEAEs | (%) u | x ( xx.x) | x (x xx )x | x ( xx.x) | x (xx x) |
| MedDRA® System Organ Class 1<br>MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | n(%)<br>n(%)<br>n(%) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x)<br>x (xx x) | x ( xx.x) x ( xx.x) x ( xx.x) x ( xx.x) x | x (xx x) x (xx x) x (xx x) x |
| MedDRA® System Organ Class 2<br>MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | n(%)<br>n(%)<br>n(%) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x)<br>x (xx x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx x)<br>x ( xx x)<br>x ( xx x) |
| MedDRA® System Organ Class 3<br>MedDRA® Preferred Term 1<br>MedDRA® Preferred Term 2 | n(%)<br>n(%)<br>n(%) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x)<br>x (xx x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x (xx x)<br>x (xx x)<br>x (xx x) |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

2) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with TEAE; MedDRA ®: Medical Dictionary for Regulatory Activities, version 23.0; TEAEs: Treatment-Emergent Adverse Events.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences.

Overall: Included results from all treatment groups.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analys is Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

Table 14.3.1-8 Frequency of Subjects Experiencing Serious Treatment-Emergent Adverse Events Summarized per Treatment

Safety Population

| Saicty repaiding | | | | | |
|---|---|---|---|---|---|
| MedDRA® System Organ Class | Ctotiotic | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | 1 mg/kg US - Avastin® IV | Overall |
| MedDRA® Preferred Term | Statistic | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| | ~ ~ ~ | ` | ` | ` | |
| Number of Subjects with TEAES | n (%) | x ( xx.x) | x (xx x) | x ( xx.x) | (XXX)X |
| MedDRA® System Organ Class 1 | n(%) | x ( xx.x) | x ( xx x) | x (xx.x) | x ( xx x) |
| MedDRA® Preferred Term 1 | n(%) | x ( xx.x) | x ( xx x) | x ( xx.x) | x ( xx x) |
| $MedDRA^{\oplus}$ Preferred T erm 2 | n(%) | x ( xx.x) | x ( xx x) | x ( xx.x) | x (xx x) |
| • | | | | | |
| MedDRA® System Organ Class 2 | (%)u | x (xx.x) | x ( xx x) | x ( xx.x) | x ( xx x) |
| MedDRA® Preferred Term 1 | n(%) | x ( xx.x) | x ( xx x) | x ( xx.x) | x ( xx x) |
| $\mathrm{MedDRA}^{\otimes}$ Preferred Term 2 | n(%) | X(XX.X) | x ( xx x) | x ( xx.x) | x ( xx x) |
| € | : | | | | |
| MedDRA® System Organ Class 3 | (%)u | x ( xx.x) | x(xx) | x ( xx.x) | x ( xx x) |
| MedDRA® Preferred Term 1 | n(%) | x ( xx.x) | x ( xx x) | x(xx.x) | x ( xx x) |
| MedDRA® Preferred Term 2 | u(%) | x ( xx.x) | x ( xx x) | x ( xx.x) | x ( xx x) |

Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

2) Refer to footnotes for additional instructions

N: Number of subjects dosed; n (%): Number and percent of subjects with TEAE; MedDRA®: Medical Dictionary for Regulatory Activities, version 23.0; TEAEs: Treatment-Emergent Adverse Events.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences.

Overall: Included results from all treatment groups.



Statistical Analysis Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Spons or Study Number: MB02-A-06-20)

| Darameter | | | | |
|---|---|---|---|---|
| alameter | | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | 1 mg/kg US - Avastin® IV |
| (unit) Visit | Statistic | (XX=N) | (N=XX) | (XX=N) |
| Parameter 1 Screening | п | XX | XX | XX |
| XX-XX | Mean | xx.x | X XX | X XX |
| | SD | XX.X | X XX | X XX |
| | Median | XX.X | X XX | X XX |
| | Min, Max | xx-xx | xx-xx | xx-xx |
| Day -1 | п | XX | XX | XX |
| | Mean | XX.X | X XX | X XX |
| | SD | XX.X | X X X | X XX |
| | Median | XX.X | X X X | X XX |
| | Min, Max | XX-XX | xx-xx | XX-XX |
| Baseline | п | XX | XX | XX |
| | Mean | XX.X | X XX | X XX |
| | S | XX.X | X XX | X XX |
| | Median | XX.X | X XX | X XX |
| | Min, Max | XX-XX | XX-XX | XX-XX |
| Day 3 | n | XX | xx | XX |
| | Mean | XX.X | X XX | X XX |
| | S | XX.X | X XX | X XX |
| | Median | XX.X | X XX | X XX |
| | Min, Max | XX-XX | XX-XX | XX-XX |
| Day3 - CFB | u | xx | xx | xx |
| | Mean | XX.X | X X X | X XX |
| | S | XX.X | X XX | X XX |
| | Median | XX.X | X XX | X XX |
| | Min, Max | XX-XX | xx-xx | XX-XX |
| Day 8 | u | xx | xx | xx |
| | Mean | XX.X | X XX | X XX |
| | S | XX.X | X XX | X XX |
| | Median | XX.X | X XX | X XX |
| | Min, Max | XX-XX | XX-XX | XX-XX |



Project Number 7012755 (Spons or Study Number: MB02-A-06-20) Statistical Analysis Plan (Table/Figure/Listing Shells)

| Table 14.3.4-1 Clinical | Chemistry Sumr | nary Descriptive Statistics | Table 14.3.4-1 Clinical Chemistry Summary Descriptive Statistics and Change from Baseline - Safety Population | Safe ty Population |
|---|---|---|---|---|
| Parameter | | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | 1 mg/kg US - Avastin®IV |
| (unit) | | (N=XX) | (N=XX) | (XX=N) |
| Visit | Statistic | | | (**** |
| Day - CFB | п | XX | xx | xx |
| | Mean | XX.X | X X X | X XX |
| | SD | XX.X | X X X | X XX |
| | Median | XX.X | X X X | X XX |
| | Min, Max | xx-xx | XX-XX | XX-XX |
| : | | | | |
| End of Study (Day 100) n | )ay 100) n | XX | xx | xx |
| | Mean | XX.X | X X X | X XX |
| | SD | XX.X | X X X | X XX |
| | Median | XX.X | X X X | X XX |
| | Min, Max | xx-xx | xx-xx | XX-XX |
| End of Study (Day 100) - n<br>CFB | )ay 100) - n | xx | xx | xx |
| | Mean | XX.X | X XX | X XX |
| | S | XX.X | X X X | X XX |
| | Median | XX.X | X X X | X XX |
| | Min, Max | XX-XX | XX-XX | XX-XX |

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to the study drug administration. CFB: Change from baseline; N: Number of subjects dosed; n: Number of subjects; SD: Standard Deviation. Data source: Listing 16.2.8-1 Note: This table will be repeated for Tables 14.3.4-3, 14.3.4-5, 14.3.4-7, 14.3.4-11 and 14.3.4-12. Please adapt title and footnotes accordingly.



Statistical Analysis Plan (Table/Figure/Listing Shells)

Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

| Table 14.3.4-2 Frequency of Subjects - Clinic | ncy of Subjects - C | Jinical ( | cal Chemistry Shifts from Baseline - Safety Population | hifts from I | 3 as e line | - Safe ty Po | pulation | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline Flag: | | Normal | | | AbnormalNCS | S | | Abnormal CS | |
| Treatment | Post-Baseline Flag: | Normal | Abnormal NCS Abnormal CS | AbnormalCS | Normal | Abnormal NCS Abnormal CS | Abnormal CS | Normal | Abnormal NCS Abnormal CS | Abnormal CS |
| Parameter (unit) | > | (%) u | n (%) | n (%) | (%) u | n (%) | (%) u | (%) u | n (%) | n (%) |
| 1 mg/kg MB02 - SP IV (N=XX) | () | | | | | | | | | |
| Parameter 1 | Day 3 | $(x \times x)$ | $(x \times x)$ | x ( xx.x) | x (xx.x) | x(xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | | $(x \times x)$ | $(x \times x)$ | x (xx.x) | (x.x.x) | x(xx.x) | $(x \times x)$ | (x.x.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 14 | $(x \times x)$ | $(x \times x)$ | x (xx.x) | (x.x.x) | x(xx.x) | $(x \times x)$ | (x.x.x) | $(x \times x)$ | $(x \times x)$ |
| | | $(x \times x)$ | $(x \times x)$ | x ( xx.x) | x (xx.x) | x(xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 28 | $(x \times x)$ | $(x \times x)$ | x ( xx.x) | x (xx.x) | x(xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 42 | $(x \times x)$ | $(x \times x)$ | x ( xx.x) | x (xx.x) | x(xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 56 | $(x \times x)$ | $(x \times x)$ | x ( xx.x) | x(xx.x) | (xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 78 | $(x \times x)$ | $(x \times x)$ | x ( xx.x) | x (xx.x) | (xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 100 (End of | (x xx ) x | $(x \times x)$ | x (xx.x) | x (xx.x) | x(xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x) \times$ | $(x \times x)$ |
| | Study) | | | | | | | | | |
| Parameter 2 | Day 3 | $(x \times x)$ | $(x \times x)$ | x (xx.x) | (x.x.x) | x(xx.x) | (x xx) | x(xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 8 | $(x \times x)$ | $(x \times x)$ | x (xx.x) | x(xx.x) | x(xx.x) | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 14 | $(x \times x)$ | $(x \times x)$ | x (xx.x) | x (xx.x) | (x.x.) | $(x \times x)$ | x (xx.x) | x (xxx) | x(xxx) |
| | : | | | | | | | | | |
| E | | | | | | | | | | |
| Add for all other I reatments | | | | | | | | | | |
| and Parameters | | | | | | | | | | |

Programming Notes:

Preserve parameters, scheduled visits and sorting defined in Summary Descriptive Statistics Table
 Refer to footnotes for additional instructions.
 Adapt Data Source to the appropriate laboratory category listing.

N: Number of subjects dosed; n: Number and percent of subjects.

Percentage based on the number of subjects having available results at baseline and at the specific post-baseline timepoint. Baseline is defined as the last results (scheduled or unscheduled) obtained prior to the study drug administration.

Data source: Listing 16.2.8-1

Note: This table will be repeated for Tables 14.3.4-4, 14.3.4-6, 14.3.4-8, and 14.3.4-13 please adapts title and footnotes accordingly.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analys is Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

| Table 14.3.4-9 Urinalysis Frequen | sis Frequency S | ummary – Cat | cy Summary – Categorical Results – Safety Population | ty Population | |
|---|---|---|---|---|---|
| Parameter (unit) | | Result | 1 mg/kg MB02 - SP IV | 1 mg/kg MB02 - DM IV | 1 mg/kg US - Avastin <sup>®</sup> IV |
| Normal Range | Visit | n (%) | (N=XX) | (N=XX) | (N=XX) |
| Parameter 1(unit) | Screening | Negative | x(xxx) | $(x \times x) \times x$ | x (xx x) |
| XX-XX | | Trace | x(xxx) | x(xx) | x(xx x) |
| | Day -1 | Negative | $(x \times x)$ | x (xx x) | x (xx x) |
| | | Trace | $(x \times x) \times (x \times x)$ | $(x \times x)$ | $(x \times x)$ |
| | Baseline | Negative | x (xx x) | x (xx x) | x (xx x) |
| | | Trace | x(xxx) | x (xx x) | x (xx x) |
| | Day 8 | Negative | x (xx x) | x (xx x) | x (xx x) |
| | | Trace | x(xxx) | x (xx x) | $(x \times x)$ |
| | Day 14 | Negative | x(xxx) | x (xx x) | $(x \times x)$ |
| | | Trace | x(xxx) | x (xx x) | x (xx x) |
| | Day 21 | Negative | x(xxx) | x (xx x) | $(x \times x)$ |
| | | Trace | x(xxx) | x (xx x) | x (xx x) |
| | : | | | | |
| | Day 100 (Endof | Negative | x (x x x) | x (xx x) | $(x \times x)$ |
| | Study) | Trace | x (xx x) | x (xx x) | $(x \times x)$ |

Programming Notes:

Evaluate if the units must be added to param etername if a numeric result was observed. Remove (units) from column header if no numeric results were observed. Urine Microscopy parameters will not presented in this table.
 Evaluate if the units must be added to parameter name if a nun 3) For each parameter nowide now.

For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of gender from demographic table.

Independently for each parameter, sort results by gradation.

Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects.

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to the study drug administration.

Percentage based on the number of subjects having available result at each timepoint, in dependently for each parameter.



Statistical Analys is Plan (Table/Figure/Listing Shells)

Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

Table 14.3.4-10 Frequency of Subjects – Urinalysis Shifts from Baseline – Categorical Results – Safety Population

| Table 14.5.4-10 Firequency of Subjects - Climarysis Sinnes moin Basenine - Caregoriea incomis | - Ofmanysis Sinits in | un Dascinic - | arcguirai ive | suits – Saic iy i opmation | ршаноп |
|---|---|---|---|---|---|
| | Baseline Flag: | Normal | nal | Abno | Abnormal |
| Treatment | Post-Baseline Flag: | Normal | Abnormal | Normal | Abnormal |
| Parameter (unit) | Visit | n (%) | n (%) | n (%) | n (%) |
| 1 mg/kg MB02 - SP IV (N=XX) | | | | | |
| Parameter 1 | Day 3 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 8 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 14 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 21 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 28 | $(x \times x)$ | x(xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 42 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 56 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 78 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 100 (End of Study) | x ( xx x) | x (xx.x) | x (xx x) | $(x \times x)$ |
| Parameter 2 | Day 3 | x (xx x) | x ( xx.x) | x ( xx x) | x ( xx x) |
| | Day 8 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 14 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 21 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 28 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 42 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 56 | $(x \times x)$ | x (xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 78 | $(x \times x)$ | x(xx.x) | $(x \times x)$ | $(x \times x)$ |
| | Day 100 (End of Study) | x ( xx x) | x (xxx) | (x xx)x | (x xx)x |
| Add for all other Treatments and Parameters | | | | | |

Programming Notes:

Preserve parameters, scheduled visits and sorting defined in Summary Descriptive Statistics Table
 Refer to footnotes for additional instructions.
 Adapt Data Source to the appropriate laboratory category listing.

Adapt Data Source to the appropriate laboratory category listing.

N: Number of subjects dosed; n: Number and percent of subjects.

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to the study drug administration.

Percentage based on the number of subjects having available results at baseline and at the specific post-baseline timepoint. Data source: Listing 16.2.8-3



Statistical Analys is Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

5. Listings

20 May 2021 (Final 1.0)



mAbxience Research S.L.

| Completion and Discontinuation Information |
|--------------------------------------------|
| ormi |
| n Inf |
| atio |
| ntinu |
| iscol |
| land |
| etion |
| nmc |
| Č |
| ects |
| -1 Sub |
| <u>-</u> |
| 7 |
| 16. |
| Listing 16.2.1-1 Subjects |

| | ntinuation Comment | XXX |
|---|---|---|
| ate of Last Contact With The Prima | Subject Discor | DD-MM-YYYY XXX |
| Completion/Discontinuation Date Date of Last Contact With The Primary Reason for | and Time Su | DD-MM-YYYYYTHH:MM |
| | Date ICF signed | |
| ) | Subject Treatment Date ICF signed | 001 1 mg/kg<br>MB02 -<br>SP IV |



Statistical Analys is Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

| Listing 1 | Listing 16.2.2-1 Protocol Deviations | | |
|-----------|--------------------------------------|----------|-----------|
| Subject | Treatment | Category | Deviation |
| | 1 mg/kg MB02 - SP IV | | |



mAbxience Research S.L.

| • |
|---|

| LISUING I | 0.2.4-1 Demo | grapmes | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | Visit | Treatment | Age (years) | Race | Ethnicity | $BMI (kg/m^2)$ | Height (cm) | Weight (kg) |
| 001 | Screening | 1 mg/kg MB02 - SP IV | | | | | | |

BMI: Body Mass Index. Last results (scheduled or unscheduled) obtained at screening were used to generate this listing.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analysis Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

## Listing 16.2.4-2 Medical History Findings at Screening

| Subject Treatment Finding MedDRA® Preferred Term MedDRA® System Organ Class Onset Date (or Ongoing) I mg/kg MB02 - SP IV FINDING 1 Preferred Term 1 SOC 1 YYYY-MM-DDTHH:MM YYYYY-MM-DDTHH:MM ONGOING | | | , | ) | | | Decolution Date |
|---|---|---|---|---|---|---|---|
| B02 - SP IV FINDING 2 Preferred Term 1 SOC 1 FINDING 2 Preferred Term 2 SOC 2 | ubject | Treatment | Finding | MedDRA® Preferred Term | MedDRA® System Organ Class | Onset Date | (or Ongoing) |
| FINDING 2 Preferred Term 2 SOC 2 | | | FINDING 1 | Preferred Term 1 | SOC 1 | YYYY-MM-DDTHH:MM | YYYY-MM-DDTHH:MM |
| FINDING 2 Preferred Term 2 SOC 2 | | 1 mg/kg MB02 - SP IV | | | | | |
| | | 1 | FINDING 2 | Preferred Term 2 | SOC 2 | YYYY-MM-DDT HH:MM | ONGOING |

Programming Notes

SOC and Finding will be presented in uppercase. The Preferred Term will be presented in "propease". The SAS coding "/~n" between terms will generate the break line.
 If The SAS coding "/~n" between dates will generate the break line.
 Iffinding is ongoing, replace missing resolution date per ONGOING.
 Sort events per Subject, Start Date, Stop Date, Stoc and PT.

5) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format. MedDRA®: Medical Dictionary for Regulatory Activities; MedDRA® Version 23.0.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analysis Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

## Listing 16.2.4-3 Prior and Concomitant Medications

| - | | | 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | | |
|---|---|---|---|---|---|---|---|
| | | | WHO DDE ATC/ | | | Onset Date and Time/ | |
| | Treatment | Prior/ | WHO DDE PreferredTerm/ | Dose (unit)/ | | Resolution Date and Time | Indication |
| Subject | | Concomitant | Medication | Frequency | Route | Route (or Ongoing) | (Condition or AE No.) |
| | | Prior | ATC1/ | 20 (mg) | ORAL | YYYY-MM-DDTHH:MM/ | |
| | | | PreferredTerm 1/ | QID | | YYYY-MM-DDT HH:MM | |
| | | | MEDICATION 1/ | | | | |
| | 1 MD0.7 .cm | , | C C H | | | WWW MM PDT HHAMM | |
| | I mg/kg Mb02 - Sr | Concomitant | AIC2/ | | | I I I I - MIM-DDI HH:MIM/ | |
| | IV | | Preferred Term 2/ | | | ONGOING | |
| | | | MEDICATION 2/ | | | | |

Programming Notes:

1) ATC and Medication will be presented in uppercase. The Preferred Term will be presented in "propoase". The SAS coding "/~n" between terms will generate the break line.

2) The SAS coding "/~n" will generate the break line between treatment sequence and treatment, dose with units and frequency. In the same way apply a break line between

If medication is ongoing, replace missing resolution date per ONGOING.
 Sort events per Subject, Onset Date, Resolution Date, ATC and PT.

5) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.

ATC: Anatomic Therapeutic Chemical; WHODDE: World Health Organization Drug Dictionary Enhanced Version Mar 2020, format B3.



Statistical Analysis Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

Listing 16.2.4-4 Study Drug Administration

| | | | | | | | | DDT HH:MM:SS | DDT HH:MM:SS | | MB02 -<br>SP IV | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | YYYY-MM- | YYYY-MM- | | 1 mg/kg | |
| interrupted? | Status | administration | (mL) | (unit) | administered? | (mg) | (hh: min) | Date and Time | Reason" Date and Time | Reason" | Subject Treatment | Subject |
| infusion | Fasting | study drug | infused | Rate | volume | Weight | infusion | Infusion End | Infusion Start | If No, | | |
| Wasthe | | Location of | | Infusion | Was the total | subject | Jo | | | Taken/ | | |
| | | | | | | Dose per | Duration | | | Drug | | |
| | | | | | | Total | | | | | | |



Statistical Analysis Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

| Drug Interruption Restart nent Date and Time Date and Time Reason for interruption sg MB02 - YYYY-MM- DDTHH-MM-SS DDTHH-MM-SS | | | | and a rest of the control of the con | LISTING TO |
|---|---|---|---|---|---|
| g MB02 - YYYY-MM- | Reason for interruption | Restart<br>Date and Time | | | Subject |
| S-MM·HHTQQ | | YYYY-MM- | | , | |
| | | DDT HH:MM:SS | SS | SP IV | |



Statistical Analysis Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

## Listing 16.2.4-6 Assignment to Analysis Populations

| Included in Safety Population | Yes |
|-------------------------------|----------------------|
| Treatment | 1 mg/kg MB02 - SP IV |
| Subject | 101 |



mAbxience Research S.L.

## Listing 16.2.4-7 Cotinine Test

| Treatment | Visit | Test Performed/ If No,<br>Reason | Date/Time of Sample<br>Collection | Result |
|---|---|---|---|---|
| 1 mg/kg MB02 -SP IV | Screening | Yes | ddmmmyyyy / hh mm | Negative |
| | Day -1 | Yes | ddmmmyyyy / hh mm | Positive |
| | Screening | No | | |
| | Day -1 | Yes | ddmmmyyyy / hh mm | Negative |



mAbxience Research S.L.

### Listing 16.2.4-8 Urine Drug Screen

| Test Name If<br>Positive Results | | | | | |
|---|---|---|---|---|---|
| Result | Negative | Positive | | Negative | |
| Date/Time of Sample<br>Collection | ddmmnyyyy / hh mm | ddmmnyyyy / hh mm | | ddmmnyyyy / hh mm | |
| Test Performed/IfNo,<br>Reason | Yes | Yes | No | Yes | |
| Visit | Screening | Day -1 | Screening | Day-1 | |
| Treatment | 1 mg/kg MB02 - SP | ≥ | | | |
| Subject | XXXXX | | XXXXX | | etc. |



mAbxience Research S.L.

## Listing 16.2.4-9 Alcohol Breath Test

| Result | Negative | Positive | | Negative | |
|---|---|---|---|---|---|
| Date/Time of Sample<br>Collection | ddmmnyyyy / hh mm | ddmmnyyyy / hh mm | | ddmmmyyyy / hh mm | |
| Test Performed/IfNo,<br>Reason | Yes | Yes | No | Yes | |
| Visit | Screening | Day-1 | Screening | Day-1 | |
| Treatment | 1 mg/kg MB02 - SP IV | | | | |
| Subject | XXXXX | | XXXXX | | etc. |



able/Figure/Listing Shells)

mAbxience Research S.L.

### Listing 16.2.4-10 Randomization

| Randomization Number. | |
|---------------------------------------|----------------------|
| Randomization Date | ddmmmyvyv |
| Subject Was Randomized / IfNo, Reason | |
| Treatment | 1 mg/kg MB02 - SP IV |
| Subject | 101 |



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analysis Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

## Listing 16.2.7-1 Non-Treatment-Emergent Adverse Events

Subject

| | MedDRA <sup>®</sup> System Organ Class/ | Onset Date and Time/ | | Other | | Action taken | ken | |
|---|---|---|---|---|---|---|---|---|
| AE Number | MedDRA® Preferred Term/<br>AE Number Adverse Event Description | Resolution Date and Time (or Ongoing) | Severity/<br>Relationship | causal Serious<br>relationship (Yes/No) | Serious<br>(Yes/No) | Study Drug Other Outcome | Other | Outcome |
| | SOC 1/<br>Preferred Term 1/<br>DESCRIPTION 1 | YYYY-MM-DDTHH:MM/<br>YYYY-MM-DDTHH:MM | Severe/<br>Unrelated | | Yes | | | |
| | SOC 2/<br>Preferred Term 2/<br>DESCRIPTION 2 | YYYY-MM-DDTHH:MM/<br>ONGOING | Mild/ | | No | | | |

Programming Notes

1) SOC and AE Description will be presented in uppercase. The Preferred Term will be presented in "propoase". The SAS coding "/-n" between terms will generate the break line.

2) The SAS coding "/-n" will generate the break line between dates and between Severity and Relationship

If needed, hardcode OUTCOME and ACTIONS in order to introduce break line (-n) between answer elements.

4) If medication is ongoing, replace missing resolution date per ONGOING.

5) Sort events per Subject, Onset Date/time, Resolution Date/time, SOC and PT.

6) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
 7) Please update' MedDRA\* System Organ Class' footnote by keeping only those SOC terms referred in table.
 MedDRA\*: Medical Dictionary for Regulatory Activities (MedDRA\*); MedDRA\* Version 23.0

Infections and infestations (Infect); Injury, poisoning and procedural complications (Inj&P); Investigations (Inv); Musculoske letal and connective tissue disorders (Musc); Nervous system MedDRA® System Organ Class (SOC): Cardiac disorders (Card); Eye disorders (Eye); Gastrointestinal disorders (Gastr); General disorders and administration site conditions (Gentl); disorders (Nerv); Psychiatric disorders (Psych); Respiratory, thoracic and mediastinal disorders (Resp); Skin and subcutaneous tissue disorders (Skin) Vascular disorders (Vasc).

Note: The list of MedDRA ® SOC will be updated according to the A Es observed for the study.



Project Number 7012755 (Sponsor Study Number: MB02-A-06-20) Statistical Analysis Plan (Table/Figure/Listing Shells)

mAbxience Research S.L.

| Listi | ng 16.2.7 | -2 Trea | Listing 16.2.7-2 Treatment-Emergent Adverse Events | se Events | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | MedDRA® System Organ | | | | | Actiontaken | aken | |
| | | AE | Class/<br>MedDRA® Preferred Term/ | Onset Date and Time/<br>Resolution Date and Time Severity/ | Severity/ | Other causal | Serions | | | I |
| Subject | Treatment | Number | Subject Treatment Number Adverse Event Description | (or Ongoing) | Relationship | relationship (Yes/No) | (Yes/No) | Study Drug Other Outcome | Other | Outcome |
| 001 | 1 mg/kg<br>MB02 - SP<br>IV | | SOC 1/<br>PreferredTerm 1/<br>DESCRIPTION 1 | YYYY-MM-DDTHH:MM/ Grade 1/<br>YYYY-MM-DDTHH:MM Unrelated | Grade 1/<br>Unrelated | | Yes | | | |
| | | | SOC 2/<br>Preferred Term 2/<br>DESCRIPTION 2 | YYYY-MM-DDTHH:MM/ Grade 2/<br>ONGOING Remote | Grade 2/<br>Remote | | No | | | |

Programming Notes:

1) SOC and AE Description will be presented in uppercase. The Preferred Term will be presented in "propcase". The SAS coding "/~n" between terms will generate the break line.

2) The SAS coding "/-n" will generate the break line between dates and between Severity and Relationship.

3) If needed, hardcode OUTCOME and ACTIONS in order to introduce break line (~n) between answer elements.

5) Sort events per Subject, Onset Date/time, Resolution Date/time, SOC and PT. 4) If medication is ongoing, replace missing resolution date per ONGOING.

6) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.

7) Please updaie' MedDR4® System Organ Class' footnote by keeping only those SOC terms referred in table. MedDRA®: Medical Dictionary for Regulatory Activities (MedDRA®); MedDRA® Version 23.0

Infections and infestations (Infec); Injury, poisoning and procedural complications (Inj&P); Investigations (Inv); Musculosk eletal and connective tissue disorders (Musc); Nervous system MedDRA® System Organ Class (SOC): Cardiac disorders (Card); Eye disorders (Eye); Gastrointestinal disorders (Gastr); General disorders and administration site conditions (Genrl); disorders (Nerv); Psy chiatric disorders (Psych); Respiratory, thoracic and mediastinal disorders (Resp); Skin and subcutaneous tissue disorders (Skin) Vascular disorders (Vasc).

Note: The list of MedDRA ® SOC will be updated according to the ABs observed for the study.

Note: Similar layout will be used for Listing 16.2.7-3, 16.2.7-4 and 16.2.7-5 please adapttitle and footnotes accordingly.



mAbxience Research S.L.

| Collection Date Collection Date Solution and Time | Subject Treatment Laboratory Visit | Collection Date | Parameter(1mit) | Norm<br>Result Result | Normalized<br>Result | NormalRange | Flao | Interpretation |
|---|---|---|---|---|---|---|---|---|
| Toman 1 | ner Cromcom | 2000 1 2000 | _ | ancour. | 12000 | Sumurane | 2 | THE DESCRIPTION |
| 1 mg/kg<br>MB02 -<br>SP IV | | YYYY-MM-<br>DDT HH:MM | | | | XX.X-XXX | Н | Abnormal NCS |

Programming Notes:

1) Sort assessments per Subject, Timepoint/Date and parameters. Sorting for parameter should be as defined in Summary Descriptive Statistics Table.
2) For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of gender from demographic table.

If multiple laboratories involved, display standard and normalised results. Display the ranges in the same way. The SAS coding "/-n" between results or ranges will generate the break line. Take care to use the same precision of both, standard and normalised results/ranges.

Laboratory facilities could be abbreviated with appropriation description on footnote; BML: Biron Medical Laboratory).

H: Above normal range; L: Below normal range; N: Normal Range.

Note: Similar layout will be used for Listings 16.2.8-2, 16.2.8-3, 16.2.8-4, 16.2.8-5, and 16.2.8-6. Please adapt title and footnotes accordingly.



Statistical Analysis Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

| Listing 16 | .2.8-7 Vital | Listing 16.2.8-7 Vital Signs Result | | | |
|---|---|---|---|---|---|
| | | Vis it/ | Measurement Date and | | |
| Subject | Subject Treatment Timepoint | | Time | Parameter(unit) | Result |
| | ! | | | | |
| 001 | 1 mg/kg<br>MB02 - SP | Screening | YYYY-MM-<br>DDTHH·MM | | |
| | <u> </u> | | | | |

Programming Notes:

1) Sort assessments per Subject, Timepoint/Date and parameter. Parameters for each subject to be sorted as defined in Summary De scriptive Statistics Table.

1) Sort assessments per Subject, Timepoint/Date and parameter. Parameters for each subject to be sorted as defined in Summary De scriptive Statistics Table.

\*The medical judgement for abnormal ECG interpretation is also presented in this column as CS: Clinically significant or NCS: Not clinically significant.



mAbxience Research S.L.

| Listing 10 | 5.2.8-8 Pulse | is ting 16.2.8-8 Pulse Oximetry Results | ults | | | |
|---|---|---|---|---|---|---|
| Subject | Subject Treatment Visit | Visit | Start Date and Time | Test (unit) | Result | Reason, if Test is Not Performed |
| 001 | 1 mg/kg<br>MB02 - SP<br>IV | Screening | ҮҮҮҮ-ММ-ДБТНН:ММ | | | |



mAbxience Research S.L.

| Listing | Listing 16.2.8-9 Electroca | ĭ | diogram Result | | | |
|---|---|---|---|---|---|---|
| Subject | Treatment | Visit/Timepoint | Assessment Date and Time | Parameter(unit) | Result | Interpretation* |
| | 1 mg/kg<br>MB02 - SP | | үүүү-мм-рртнн:мм | | | |

 $\geq$ 

Programming Notes:

Note: Similar layout will be used for Listings 16.2.8-10, and 16.2.8-11. Please adapt title and footnotes accordingly

<sup>1)</sup> Sort assessments per Subject, timepoint/Date and parameter: Parameters for each subject to be sorted as defined in Summary Descriptive Statistics Table.

\*The medical judgement for abnormal ECG interpretation is also presented in this column as CS. Clinically significant or NCS. Not clinically significant.



Statistical Analysis Plan (Table/Figure/Listing Shells)
Project Number 7012755 (Sponsor Study Number: MB02-A-06-20)

| | Treatment | Timepoint | Examination Date and Time | Sit e/System | Results |
|---|---|---|---|---|---|
| 101/29 | 1 mg/kg MB02 - SP IV | Screening | YYYY-MM-DDTHH:MM | General Appearance | Normal |
| | | | | Eye/Ear/Nose/Throat | Normal |
| | | | | Oral | Normal |
| | | | | Head and Neck | Normal |
| | | | | Chest/Lungs | Normal |
| | | | | Abdomen | Normal |
| | | | | Lymphatic | Normal |
| | | | | Neurologic | Normal |
| | | | | Extremities | NE |
| | | | | Psychiatric | NE |
| | | | | Other | NE |

NE: not evaluated.